CLINICAL TRIAL: NCT00740116
Title: Tranexamic Acid in Surgery of Advanced Ovarian Cancer - a Prospective Randomized Double Blind Placebo Controlled Study
Brief Title: Tranexamic Acid in Surgery of Advanced Ovarian Cancer
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Preben Kjolhede, MD, professor (Other)
Responsible Party: Sponsor-Investigator, Preben Kjolhede, MD, professor, Associate professor, University Hospital, Linkoeping
Organization: University Hospital, Linkoeping (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EudraCT nr 2006-006714-14
Record Dates: First submitted 2008-08-21; First posted 2008-08-22 (Estimated); Results first posted 2022-03-15 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-01

CONDITIONS: Ovarian Cancer
Keywords: Tumor of ovary; Surgical blood loss; Postoperative blood loss; Preventive therapy; Thromboembolism
MeSH Terms: conditions — Ovarian Neoplasms; Blood Loss, Surgical; Postoperative Hemorrhage; Thromboembolism | interventions — Tranexamic Acid; Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- The Tranexamic acid group (Active Comparator): The group of women receiving Tranexamic acid intravenously immediately before the surgery
  Interventions: Drug: Tranexamic acid
- The placebo group (Placebo Comparator): The group of women receiving saline solution (0.9% NaCl) intravenously immediately before the surgery
  Interventions: Drug: 0.9% NaCl solution

INTERVENTIONS:
Drug: Tranexamic acid — Tranexamic acid, 100 mg/ml; 15 mg/kg body weight added to 100 ml 0.9% NaCl solution given as a single dose intravenously immediately prior to skin incision at surgery
  Other Names: Cyklokapron; ATC-code B02AA02
  Arms: The Tranexamic acid group
Drug: 0.9% NaCl solution — 0.9% NaCl solution; 0.15 ml/kg body weight added to 100 ml 0.9% NaCl solution. The volume is given intravenously immediate before skin incision at surgery.
  Other Names: 0.9 % sodium chloride; ATC-code B05BB01
  Arms: The placebo group

SUMMARY:
The purpose of the study is to determine if a standardized single dose tranexamic acid given intravenously immediately preoperatively reduces the perioperative bleeding volume and reduces the need of blood transfusion in women undergoing surgery for advanced ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

* Females ages 18 or older with a pelvic or abdominal tumor suspected or histopathologically proven ovarian cancer FIGO stage II-IV who are undergoing primary surgery with the intention of performing optimal cytoreductive radical surgery.
* Understand and speak Swedish
* Accept participation in the study after written and verbal information and sign informed consent.

Exclusion Criteria:

* Allergy to tranexamic acid
* Having had tranexamic acid within the recent 30 days
* Previous or present episode of thromboembolic events .
* Previous or present treatment within the recent 3 months with anticoagulant.
* Previous or present known coagulopathy
* Myocardial infarction within the previous 12 months or instable angina pectoris which, according to the investigator, may increase the risk for complications significantly in case of a lowering of the hemoglobin.
* Significant renal failure with serum-creatinine > 250 µmol/l.
* Severe psychiatric dysfunction or mentally substantially disabled.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2008-03; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ulf Leandersson, MD, Principal Investigator — Dept. of Obstetrics and Gynecology, Kalmar Central Hospital, 391 85 Kalmar; Laila Falknäs, MD, Principal Investigator — Dept of Obstetrics and Gynecology, Ryhov Central Hospital, 58185 Jönköping; Preben Kjölhede, MD,PhD, Study Chair — Department of Obstetrics and Gynecology, University Hospital, Linköping; Torsten Johansson, MD, PhD, Study Chair — Dept. of Orthopedic Surgery, University Hospital, 58185 Linköping Sweden; Helena Zachrisson, MD,PhD, Study Chair — Dept of Physiology, University Hospital, 58185 Linköping Sweden
Locations (3):
- Sweden (3):
  - Dept of Obstetric and Gynecology, Ryhov Central Hospital, Jönköping
  - Department of Obstetrics and Gynecology, Kalmar Central Hospital, Kalmar
  - University Hospital, Department of Obsterics and Gynecology,, Linköping

REFERENCES:
- [Background] Nielsen HJ. Detrimental effects of perioperative blood transfusion. Br J Surg. 1995 May;82(5):582-7. doi: 10.1002/bjs.1800820505. PMID 7613921
- [Background] Lindoff C, Rybo G, Astedt B. Treatment with tranexamic acid during pregnancy, and the risk of thrombo-embolic complications. Thromb Haemost. 1993 Aug 2;70(2):238-40. PMID 8236125
- [Background] Dunn CJ, Goa KL. Tranexamic acid: a review of its use in surgery and other indications. Drugs. 1999 Jun;57(6):1005-32. doi: 10.2165/00003495-199957060-00017. PMID 10400410
- [Background] Gai MY, Wu LF, Su QF, Tatsumoto K. Clinical observation of blood loss reduced by tranexamic acid during and after caesarian section: a multi-center, randomized trial. Eur J Obstet Gynecol Reprod Biol. 2004 Feb 10;112(2):154-7. doi: 10.1016/s0301-2115(03)00287-2. PMID 14746950
- [Background] Johansson T, Pettersson LG, Lisander B. Tranexamic acid in total hip arthroplasty saves blood and money: a randomized, double-blind study in 100 patients. Acta Orthop. 2005 Jun;76(3):314-9. PMID 16156456
- [Background] Abu-Rustum NR, Richard S, Wilton A, Lev G, Sonoda Y, Hensley ML, Gemignani M, Barakat RR, Chi DS. Transfusion utilization during adnexal or peritoneal cancer surgery: effects on symptomatic venous thromboembolism and survival. Gynecol Oncol. 2005 Nov;99(2):320-6. doi: 10.1016/j.ygyno.2005.06.017. Epub 2005 Aug 2. PMID 16061278
- [Background] Nadler SB, Hidalgo JH, Bloch T. Prediction of blood volume in normal human adults. Surgery. 1962 Feb;51(2):224-32. No abstract available. PMID 21936146
- [Background] Brecher ME, Monk T, Goodnough LT. A standardized method for calculating blood loss. Transfusion. 1997 Oct;37(10):1070-4. doi: 10.1046/j.1537-2995.1997.371098016448.x. PMID 9354828
- [Background] Johansson T, Lisander B, Ivarsson I. Mild hypothermia does not increase blood loss during total hip arthroplasty. Acta Anaesthesiol Scand. 1999 Nov;43(10):1005-10. doi: 10.1034/j.1399-6576.1999.431006.x. PMID 10593462
- [Background] Zohar E, Fredman B, Ellis MH, Ifrach N, Stern A, Jedeikin R. A comparative study of the postoperative allogeneic blood-sparing effects of tranexamic acid and of desmopressin after total knee replacement. Transfusion. 2001 Oct;41(10):1285-9. doi: 10.1046/j.1537-2995.2001.41101285.x. PMID 11606830
- [Background] Dolan S, Fitch M. The management of venous thromboembolism in cancer patients. Br J Nurs. 2007 Nov 22-Dec 12;16(21):1308-12. doi: 10.12968/bjon.2007.16.21.27715. PMID 18073666

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between March 2008 and May 2012 one hundred women with presumed advanced ovarian cancer scheduled for radical debulking surgery att one of two university hospitals or two central hospitals in the southeast health region of Sweden and who complied with inclusion/exclusion criteria were asked to participate in the study.
Pre-assignment Details: No significant events occured after participant enrollment prior to assignment to a group.
Groups:
- Tranexamic Group: Tranexamic acid
  Tranexamic acid: Tranexamic acid, 100 mg/ml; 15 mg/kg body weight added to 100 ml 0.9% NaCl solution given as a single dose intravenously immediately prior to scin incision at surgery
- Placebo Group: 0.9% NaCl solution
  0.9% NaCl solution: 0.9% NaCl solution; 0.15 ml/kg body weight added to 100 ml 0.9% NaCl solution. The volume is given intravenously immediate before scin incision at surgery.
Period: Overall Study
Arm/Group | Tranexamic Group | Placebo Group
Started | 50 | 50
Completed | 48 | 45
Not Completed | 2 | 5
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Protocol Violation | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tranexamic Group | Placebo Group | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Continuous [Median (Full Range); unit: years] | 63 [33 to 82] | 64.5 [46 to 90] | 63 [33 to 90]
Age, Customized [Number; unit: participants]
  <60 years of age | 15 | 15 | 30
  60-69 years of age | 24 | 17 | 41
  >=70 years of age | 11 | 18 | 29
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 50 | 50 | 100
Region of Enrollment [Number; unit: participants]
  Sweden | 50 | 50 | 100
Height [Median (Full Range); unit: meter] | 1.67 [1.54 to 1.78] | 1.63 [1.45 to 1.74] | 1.64 [1.45 to 1.78]
Weight [Median (Full Range); unit: kilogram] | 71 [45.9 to 106.3] | 64.3 [46 to 117] | 67.6 [45.9 to 117]
Body mass index [Median (Full Range); unit: kg/m^2] | 25.9 [17.9 to 35.2] | 24 [16.7 to 43.5] | 25.1 [16.7 to 43.5]
Body mass index [Number; unit: participants]
  Normal weight (BMI<25) | 19 | 31 | 50
  Overweight (BMI 25-29) | 25 | 14 | 39
  Obese (BMI >=30) | 6 | 5 | 11
Parity [Median (Full Range); unit: births] | 2 [0 to 4] | 2 [0 to 5] | 2 [0 to 5]
Smokers [Number; unit: participants] | 8 | 5 | 13
Low-dose aspirin medication [Number; unit: participants] | 7 | 5 | 12
Cardiac disease [Number; unit: participants] | 5 | 1 | 6
Arterial hypertension/vascular disease [Number; unit: participants] | 22 | 13 | 35
Diabetes mellitus [Number; unit: participants] | 3 | 7 | 10
Previous hysterectomy [Number; unit: participants] | 6 | 3 | 9
Previous laparotomy [Number; unit: participants] | 25 | 21 | 46
Predicted Blood Volume (PBV) [Median (Full Range); unit: liter] | 4.16 [3.16 to 5.71] | 3.87 [2.9 to 5.71] | 3.99 [2.9 to 5.71]
RBC transfusion preoperatively [Number; unit: participants] | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Perioperative Bleeding Volume
Description: Estimation of total blood loss was based on the estimation of the Hb balance method (Brecher, et al.1997) with the assumption that the body blood volume was normalised on the fifth postoperative day. The haemoglobin level was assessed preoperatively and on the fifth postoperative day. The predicted blood volume (PBV, l) was calculated according to the method described by Nadler et al. (1962), using body weight and height. The extravasation of haemoglobin was calculated taking into account allogenic transfused haemoglobin. Total blood loss perioperatively was related to the patient's preoperative haemoglobin value. Blood loss due to haematomas or a reoperation within the first five days after surgery was also considered.
Time Frame: From start of operation to discharge from hospital, up to 5 weeks
Population: All patients underwent surgery. A negative value of total blood loss was received when the postoperative haemoglobin level was higher than the preoperative haemoglobin or when a blood transfusion was given, based on the Hb balance method of blood loss calculation.
Measure: Median (Full Range); unit: milliliter
Arm/Group | Tranexamic Group | Placebo Group
Number analyzed (Participants) | 50 | 50
milliliter | 520 [-772 to 3351] | 730 [23 to 3855]
Statistical Analysis 1: Comparison: Tranexamic Group vs Placebo Group; Test type: Superiority; p = 0.03, Wilcoxon (Mann-Whitney) — Statistical significance threshold was p < 0.05; Mann-Whitney U-test, one-sided test

2. Secondary Outcome: Number of Patients Receiving Blood Transfusions
Description: Total number of RBC-transfused women in each group
Time Frame: From start of operation to discharge from hospital, up to 5 weeks
Measure: Number; unit: participants
Arm/Group | Tranexamic Group | Placebo Group
Number analyzed (Participants) | 50 | 50
participants | 15 | 22
Statistical Analysis 1: Comparison: Tranexamic Group vs Placebo Group; Test type: Superiority; p = 0.07, Wilcoxon (Mann-Whitney) — Statistical significance threshold was p < 0.05; Mann-Whitney U-test, one-sided test

3. Secondary Outcome: Number of Units of Red Blood Cells (RBC) Transfused
Description: Total number of red blood cells (RBC) transfused across all participants
Time Frame: From start of operation to discharge from hospital, up to 5 weeks
Measure: Number; unit: units
Arm/Group | Tranexamic Group | Placebo Group
Number analyzed (Participants) | 50 | 50
units | 38 | 53
Statistical Analysis 1: Comparison: Tranexamic Group vs Placebo Group; Test type: Superiority; p = 0.46, Wilcoxon (Mann-Whitney) — Statistical significance threshold was p < 0.05; Mann-Whitney U-test, one-sided test; Odds Ratio (OR) = 0.44, 95% CI 1-sided [upper limit 0.97]

4. Secondary Outcome: Median Number of Transfused Units of Red Blood Cells (RBC)
Description: Median number of red blood cells transfused among those who received RBC transfusions
Time Frame: From start of operation to discharge from hospital, up to 5 weeks
Population: Participants who received RBC transfusions
Measure: Median (Full Range); unit: units
Arm/Group | The Placebo Group | The Tranexamic Acid Group
Number analyzed (Participants) | 22 | 15
units | 2 [1 to 6] | 2 [1 to 7]
Statistical Analysis 1: Comparison: The Placebo Group vs The Tranexamic Acid Group; Test type: Superiority; p = 0.46, Wilcoxon (Mann-Whitney) — p< 0.05 for statistical significance

5. Secondary Outcome: Number of Patients With Clinically or Radiologically Verified Thromboembolic Events Within 5 Weeks Postoperatively
Description: Thromboembolic events including arterial thrombosis, muscle vein thrombosis, superficial and deep venous thrombosis.
Time Frame: From time of operation to 5 weeks postoperatively.
Population: Information about postoperative events after discharge retrieved in patient file for the patients with withdrew consent prior to 5-weeks follow-up.
  56% of the patients underwent lower extremity duplex ultrasound.
Measure: Count of Participants; unit: Participants
Arm/Group | Tranexamic Group | Placebo Group
Number analyzed (Participants) | 50 | 50
Participants | 2 | 5
Statistical Analysis 1: Comparison: Tranexamic Group vs Placebo Group; Test type: Superiority; p = 0.22, Fisher Exact — Statistical significance threshold p-value < 0.05; Odds Ratio (OR) = 0.36, 95% CI 2-sided [0.05 to 2.72]

ADVERSE EVENTS:
Time Frame: Data were collected until five weeks after surgery.
Description: Systematic and non-systematic assessment.
Arm/Group | Tranexamic Group | Placebo Group
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 10/50 | 14/50
Other Adverse Events (participants affected / at risk) | 18/50 | 17/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tranexamic Group (N=50) | Placebo Group (N=50)
Re-operations (Surgical and medical procedures) | 5 (6) | 6 (6)
Thromboembolic events (Vascular disorders) | 2 (2) | 5 (5)
Postoperative infections (Infections and infestations) | 3 (3) | 3 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tranexamic Group (N=50) | Placebo Group (N=50)
Readmissions (General disorders) | 11 (11) | 4 (4)
Postoperative infections (Infections and infestations) | 7 (7) | 13 (13)

LIMITATIONS AND CAVEATS:
The study was not powered for postoperative complications in general. Only 56% of the women participated in the duplex ultrasound assessment of the legs, which was an optional investigation according to the trial protocol. This indicates a risk of bias for the outcome of thromboembolic complications.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No